CLINICAL TRIAL: NCT01453283
Title: A Phase I Trial and Pharmacokinetic Study of Trabectedin (YONDELIS [R], ET-743) in Children and Adolescents With Relapsed or Refractory Solid Tumors
Brief Title: Tabectedin to Treat Children and Adolescents With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Brigitte C. Widemann, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070054; 07-C-0054; NCT00437047 (obsolete NCT alias)
Record Dates: First submitted 2011-10-01; First posted 2011-10-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-04

CONDITIONS: Solid Tumors
Keywords: DNA Repair; Nucleotide Excision Repair; Trabectedine; Phase I; Sarcoma; Cytotoxic; Chemotherapy; Solid Tumor; Malignant Tumor; Rhabdomyosarcoma; Ewing Sarcoma; Neuroblastoma; Wilm's Tumor; Hepatic Tumor; Brain Tumor
MeSH Terms: conditions — Sarcoma; Neoplasms; Rhabdomyosarcoma; Sarcoma, Ewing; Neuroblastoma; Wilms Tumor; Carcinoma, Hepatocellular; Brain Neoplasms | interventions — Trabectedin

INTERVENTIONS:
Drug: Trabectedin (ecteinascidin-743, ET-743, YONDELIS [R])

SUMMARY:
Background:

* Trabectedin is an experimental drug that kills some cancer cells in the laboratory and in mice by interfering with genetic material (DNA) in cancer cells.
* In some adult patients with cancer who received trabectedin, tumors grew slower or shrank.

Objectives:

* To determine a dose of trabectedin that can be given safely to children and adolescents as a 24-hour continuous infusion through a vein.
* To determine the side effects of trabectedin in children and adolescents.
* To study how the body handles trabectedin by measuring the amount of the drug in the bloodstream over time after a dose is given.
* To measure the effect of trabectedin on DNA in white blood cells.
* To determine if an individual's tumor cells have a specific proteins involved in DNA repair and if a pattern of genes can be identified in tumor samples that might help explain why trabectedin reduces tumors in some individuals and not others.
* To study genetic factors that may influence the way the body handles trabectedin.
* To see if trabectedin is beneficial in certain types of cancer.

Eligibility:

-Children between 4 year and 17 years of age with tumors that recur or no longer respond to standard treatment.

Design:

* Patients receive trabectedin as a 24-hour continuous infusion repeated every 21 days. The first three children entering the study receive a dose of 1.1 mg/m2. Subsequent groups of up to six patients receive higher doses (1.5 mg/m2 and 1.7 mg/m2) as long as the preceding dose is well tolerated. Patients enrolled at the lowest dose level may have their dose increased to the next level if they tolerated the lower dose well. Treatment may continue as long as the cancer does not worsen and the treatment is tolerated.
* Patients have blood drawn on days 1, 2, 3, 4, 5 and 7 of the first treatment cycle to study how the body handles trabectedin.
* A tumor sample obtained from a prior surgery or biopsy is examined for proteins involved in DNA repair.
* A blood sample is drawn to look for genetic factors that may influence how the body handles trabectedin.
* Patients have periodic physical examinations and blood tests. MRI or CT scans are done before starting therapy and after every two treatment cycles to evaluate the tumor.

DETAILED DESCRIPTION:
Background:

Trabectedin (ET-743) is a natural product derived from the marine tunicate Ecteinascidia turbinata. It binds to the minor groove of DNA and interacts with various transcription factors resulting in cell cycle arrest. It also inhibits transcription coupled nucleotide excision repair system inducing lethal DNA strand breaks.

In preclinical and clinical studies, trabectedin has been found to be active in many soft tissue sarcomas including leiomyosarcoma, synovial cell sarcoma, neuroblastoma, rhabdomyosarcoma, melanoma, breast, ovarian, non-small cell lung, renal and prostate carcinoma.

In adult phase I and phase II studies, trabectedin has been well-tolerated up to dose levels of 1.9mg/m(2)/dose with the most common toxicities being fatigue, neutropenia, and reversible transaminase elevations. Objective responses were seen at doses equal to or greater than 1.5mg/m(2)/dose. Trabectedin 1.5mg/m(2) administered as a 24-hour continuous intravenous infusion is the recommended dose and schedule in adults.

A pediatric phase I study of trabectedin administered as a 3-hour infusion has been completed in the Children's Oncology Group. The maximum tolerated dose was 1.1 mg/m(2). Dose limiting toxicity was reversible elevation of hepatic transaminases.

Objectives:

Determine the maximum tolerated dose (MTD) of trabectedin administered as a 24-hour continuous infusion in children and adolescents with relapsed or refractory solid tumors.

Define the toxicity profile of trabectedin administered as a 24-hr infusion in children and adolescents.

Describe the pharmacokinetics of trabectedin administered as a 24-hr infusion in children and adolescents.

Quantify double strand DNA breaks in peripheral blood mononuclear cells of patients receiving trabectedin.

Evaluate archival formalin fixed paraffin embedded tumor tissue, when available from prior biopsies or surgical procedures, for the expression of the nucleotide excision repair proteins and genomic instability markers (histone gamma-H2AX, phospho-ATM, phospho-Chk2) by immunohistochemistry

Molecular characterization of DNA repair genes and correlation to outcome using mRNA isolated from microdissected archival formalin fixed, paraffin embedded tumor sections.

Study the pharmacogenetics of host DNA repair proteins and drug metabolizing enzymes to explore the impact of host factors on trabectedin toxicity.

Eligibility:

Children greater than or equal to 4 years and less than 17 years of age with relapsed or refractory solid tumors.

Design:

Patients will receive trabectedin as a 24-hour continuous infusion repeated every 21 days. The starting dose level is 1.1mg/m(2)/dose with escalations to 1.5mg/m(2)/dose and 1.7mg/m(2)/dose.

All patients will receive dexamethasone pretreatment and growth factor support with filgrastim or pegfilgrastim.

The definition of dose-limiting hepatic toxicity will be identical to the definition used in phase I trials in adults on the same dosing schedule.

Pharmacokinetic analysis will be performed on days 1, 2, 3, 4, 5 and 7 of the first treatment cycle.

Three to six patients will be enrolled at the first dose level and up to 6 patients will be enrolled on subsequent dose levels. Dose escalation will be based on tolerability of trabectedin at the prior dose level. For patients enrolled at dose level 1 (1.1mg/m(2)), intrapatient dose escalation to dose level 2 (1.5mg/m(2)) will be allowed with subsequent cycles if no dose limiting toxicities occurred at the lower dose level. Total accrual will be up to 24 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

AGE: greater than or equal to 4 years and less than 17 years of age.

DIAGNOSIS: Histologically confirmed solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing's sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, germ cell tumors, and brain tumors with the exception that histologic confirmation is not required for patients with optic or brainstem gliomas.

MEASURABLE/EVALUABLE DISEASE: Patients must have measurable or evaluable disease.

PRIOR THERAPY: The patient's cancer must have relapsed after or failed to respond to frontline curative therapy and there must not be other potentially curative treatment options available.

* Patients must have fully recovered to less than or equal to grade 1 from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks prior to study entry.
* Growth factors: The last dose of growth factors such as filgrastim and epoetin must be at least one week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be 2 weeks prior to study entry.
* Investigational anti-cancer agents: The last dose of all investigational agents must be at least 30 days prior to study entry.
* Biologic anti-cancer agents: The last dose of non-myelosuppressive biologic agents for the treatment of the patient's cancer (example, retinoids) must be at least 7 days prior to study entry.
* Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry, TBI and craniospinal radiation must be completed at least 4 months prior to study entry. The last dose of all other local palliative radiation must be at least 2 weeks prior to study entry.
* Stem Cell Transplantation. Patients must be at least 2 months post-autologous transplant and recovered from treatment-related toxicities. Patients who have received an allogeneic transplant are excluded.

CONCOMITANT MEDICATIONS:

-Patients with brain tumors must be on a stable or tapering dose of corticosteroids for 7 days prior to the date of the baseline scan performed for the purpose of assessing response to therapy on this study.

PERFORMANCE STATUS: Patients must have a Lansky (less than or equal to 10 years old) or Karnofsky (greater than 10 years old) score of greater than or equal to 60%.

HEMATOLOGIC FUNCTION: Peripheral absolute neutrophil count greater than or equal to 1,500/microliter and a platelet count greater than or equal to 75,000/microliter independent of transfusion, and a hemoglobin of greater than or equal to 8 gm/dl (transfusion permitted to achieve this level).

HEPATIC FUNCTION:

* ALT (SGPT) and AST (SGOT) must be less than or equal to 2.5 x the upper limit of normal (ULN).
* Bilirubin must be less than or equal to ULN. If the patient has Gilbert's syndrome, normal bilirubin is not required but should be discussed with the PI or study chair.
* Alkaline phosphatase must be less than or equal to ULN for age and sex or if alkaline phosphatase greater than ULN then 5' nucleotidase must be less than or equal to ULN or the gamma-glutamyl transpeptidase (GGT) must be less than or equal to 2.5 times the ULN to be eligible.

Normal Values for Alkaline Phosphatase at the NIH Clinical Center (U/L):

Age between 4 to 6 years with a normal value (U/L) in Males 93 to 309 and a normal value (U/L) in Females 96 to 297.

Age between 7 to 9 years with a normal value (U/L) in Males 86 to 315 and a normal value (U/L) in Females 69 to 325.

Age between 10 to 12 years with a normal value (U/L) in Males 42 to 362 and a normal value (U/L) in Females 51 to 332.

Age between 13 to 15 years with a normal value (U/L) in Males 74 to 390 and a normal value (U/L) in Females 50 to 162.

Age between 16 to 18 years with a normal value (U/L) in Males 52 to 171 and a normal value (U/L) in Females 47 to 119.

OTHER: creatine kinase less than or equal to 2.5 times the ULN.

RENAL FUNCTION: Age-adjusted serum creatinine OR a creatinine clearance greater than or equal to 60 mL/min/1.73 m(2).

Age less than or equal to 5 with a serum creatinine less than or equal to 0.8 (mg/dl).

Age greater than 5 years and less than or equal to 10 with a serum creatinine of less than or equal to 1.0 (mg/dl).

Age greater than 10 and less than or equal to 15 with a serum creatinine less than or equal to 1.2 (mg/dl).

Age greater than 15 with a serum creatinine less than or equal to 1.5 (mg/dl).

EXCLUSION CRITERIA:

Patients with severe uncontrolled infections or other unrelated systemic illnesses, which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate trabectedin or are likely to interfere with the study procedures or results.

Patients with known history of xeroderma pigmentosum or other diseases with reduced DNA repair.

Pregnant or breast-feeding females. Sexually active patients must be willing to use an effective form of birth control.

Patients currently receiving other investigational agents.

Patients who have received allogeneic stem cell transplants.

Patients who have had prior therapy with trabectedin (ET-743, Yondelis).

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2006-12-20; Primary Completion 2011-10-11 (Actual); Study Completion 2011-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Fine, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gillet LC, Scharer OD. Molecular mechanisms of mammalian global genome nucleotide excision repair. Chem Rev. 2006 Feb;106(2):253-76. doi: 10.1021/cr040483f. No abstract available. PMID 16464005
- [Background] Suk R, Gurubhagavatula S, Park S, Zhou W, Su L, Lynch TJ, Wain JC, Neuberg D, Liu G, Christiani DC. Polymorphisms in ERCC1 and grade 3 or 4 toxicity in non-small cell lung cancer patients. Clin Cancer Res. 2005 Feb 15;11(4):1534-8. doi: 10.1158/1078-0432.CCR-04-1953. PMID 15746057
- [Background] Aune GJ, Furuta T, Pommier Y. Ecteinascidin 743: a novel anticancer drug with a unique mechanism of action. Anticancer Drugs. 2002 Jul;13(6):545-55. doi: 10.1097/00001813-200207000-00001. PMID 12172500